CLINICAL TRIAL: NCT04236518
Title: Nutritional Transitions to More Plant Proteins and Less Animal Proteins: Understanding the Induced Metabolic Reorientations and Searching for Their Biomarkers
Brief Title: Nutritional Transitions to More Plant Proteins and Less Animal Proteins: Understanding the Induced Metabolic Reorientations and Searching for Their Biomarkers (ProVegOmics)
Acronym: ProVegOmics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: UMR 1019, Unité de Nutrition Humaine, INRA, Centre Auvergne-Rhône Alpes (Unknown); UMR 0914, Physiologie de la Nutrition et du Comportement Alimentaire, AgroParistech (adresse si besoin: 16 rue Claude Bernard, 75231 Paris Cedex 05). (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RBHP 2019 PICKERING 2; 2019-A02447-50 (Other: ANSM)
Record Dates: First submitted 2020-01-06; First posted 2020-01-22 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Metabolic Syndrome; Hypertriglyceridemia; Fasting Blood Sugar Above Normal; Lower Than Standard HDL-cholesterol Level; Slightly Elevated Blood Pressure
Keywords: Metabolomics; Plant Proteins, Dietary; Meat Proteins; Dietary Proteins; Metabolic Syndrome; Hypertriglyceridemia; Waist Circumference
MeSH Terms: conditions — Metabolic Syndrome; Hypertriglyceridemia | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertriglyceridimic/blood sugar/HDLcholesterol/blood pressure waist phenotype/animal protein source (Experimental): 20 men or postmenopausal women between 25 and 55 years old with a high waist circumference and at the choice, one of the following criteria high triglyceridemia, blood sugar above standards,a lower than standard HDL-cholesterol level,slightly elevated blood pressure receiving diets with predominantly animal protein sources
  Interventions: Behavioral: Diets with either predominantly animal protein sources.
- Hypertriglyceridimic/blood sugar/HDLcholesterol/blood pressure waist phenotype/plant protein source (Experimental): 20 men or postmenopausal women between 25 and 55 years old with a high waist circumference and at the choice, one of the following criteria high triglyceridemia, blood sugar above standards,a lower than standard HDL-cholesterol level,slightly elevated blood pressure receiving diets with predominantly plant protein sources
  Interventions: Behavioral: Diets with predominantly plant protein sources

INTERVENTIONS:
Behavioral: Diets with either predominantly animal protein sources. — 20 men or postmenopausal women will follow for 4 weeks a controlled diet with a protein fraction constituted mainly from animal sources. At the end of the intervention period, a post-prandial exploration will be conducted with the administration of a high-fat, high-sugar meal and subsequent blood and urine sampling.
  Arms: Hypertriglyceridimic/blood sugar/HDLcholesterol/blood pressure waist phenotype/animal protein source
Behavioral: Diets with predominantly plant protein sources — 20 men or postmenopausal women will follow for 4 weeks a controlled diet with a protein fraction constituted mainly from vegetal sources. At the end of the intervention period, a post-prandial exploration will be conducted with the administration of a high-fat, high-sugar meal and subsequent blood and urine sampling.
  Arms: Hypertriglyceridimic/blood sugar/HDLcholesterol/blood pressure waist phenotype/plant protein source

SUMMARY:
The dietary shift from animal to plant protein sources is one of the key aspects of the nutritional transition towards more sustainable food system and diets. However the metabolic implication of this shift in protein sources are still poorly understood.

This project aims to characterize and understand the metabolic orientations specifically induced by animal and vegetable dietary proteins, in order to better analyze the metabolic reorientations that would result from the expected increase in the share of plant proteins in different dietary contexts, especially those of the Western type, often associated with the development of metabolic deregulations (obesity and cardiometabolic risk).

DETAILED DESCRIPTION:
The main objectives of this project are:

* Characterize the metabolic adaptations induced by animal or plant protein diets and their repercussions in terms of physiology and health.
* Characterize the medium-term metabolomic signatures induced by this shift in dietary protein sources
* Validate, in a human population, biomarkers of dietary animal or plant proteins, previously identified in pre-clinical studies.

This clinical trial is open, monocentric, controlled, randomized, with a cross experimental design.

20 men or postmenopausal women will follow for 4 weeks a controlled diet with a protein fraction constituted mainly from animal or vegetal sources. After a 2-week washout period(+21D/-7D), they will follow another 4 week of controlled diet with predominantly animal or plant protein depending on 1st intervention period diet.

At the end of each intervention period, a post-prandial exploration will be conducted with the administration of a high-fat, high-sugar meal and subsequent blood and urine sampling.

The order in which participants will received the two diets will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 35 kh/m² (terminals included)
* Waist circumference ≥ 94 cm for men and ≥80 cm for women
* at the choice, one of the following criteria: Triglyceridemia > 1.49g/L, fasting blood glucose≥ 5.6 mmol/L , a HDL cholesterol <1.03mmol/L for men or <1.29 mmol/L for women , systolic blood pressure≥ 130 mmHg or diastolic≥ 85 mmHg .

Exclusion Criteria:

* Systolic blood pressure > 150mmHg or diastolic blood pressure > 90mmHg
* pathology and medical treatment
* diabetes
* Smoking > 4 cigarettes /day
* Alcohol consumption > 2 glasses/day
* Antibiotics taken during the last 3 months before the clinical trial
* Specific diets

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
changes of blood metabolomics | day 0
  the plasma metabolome will be determined by Liquid Chromatography - Mass Spectrometry
changes of blood metabolomics | day 14
  the plasma metabolome will be determined by Liquid Chromatography - Mass Spectrometry
changes of blood metabolomics | day 28
  the plasma metabolome will be determined by Liquid Chromatography - Mass Spectrometry
changes of blood metabolomics | day 29
  the plasma metabolome will be determined by Liquid Chromatography - Mass Spectrometry
changes of blood metabolomics | day 42
  the plasma metabolome will be determined by Liquid Chromatography - Mass Spectrometry
changes of blood metabolomics | day 56
  the plasma metabolome will be determined by Liquid Chromatography - Mass Spectrometry
changes of blood metabolomics | day 70
  the plasma metabolome will be determined by Liquid Chromatography - Mass Spectrometry
changes of blood metabolomics | day 71
  the plasma metabolome will be determined by Liquid Chromatography - Mass Spectrometry

SECONDARY OUTCOMES:
Changes of urine metabolomics | day 0
  the urine metabolome will be determined by Liquid Chromatography - Mass Spectrometry
Changes of urine metabolomics | day 14
  the urine metabolome will be determined by Liquid Chromatography - Mass Spectrometry
Changes of urine metabolomics | day 28
  the urine metabolome will be determined by Liquid Chromatography - Mass Spectrometry
Changes of urine metabolomics | day 29
  the urine metabolome will be determined by Liquid Chromatography - Mass Spectrometry
Changes of urine metabolomics | day 42
  the urine metabolome will be determined by Liquid Chromatography - Mass Spectrometry
Changes of urine metabolomics | day 56
  the urine metabolome will be determined by Liquid Chromatography - Mass Spectrometry
Changes of urine metabolomics | day 70
  the urine metabolome will be determined by Liquid Chromatography - Mass Spectrometry
Changes of urine metabolomics | day 71
  the urine metabolome will be determined by Liquid Chromatography - Mass Spectrometry
Changes in blood glucose | day 0
  The glucose concentrations will be determined by the blood samples taken by ELISA
Changes in blood glucose | day 14
  The glucose concentrations will be determined by the blood samples taken by ELISA
Changes in blood glucose | day 28
  The glucose concentrations will be determined by the blood samples taken by ELISA
Changes in blood glucose | day 29
  The glucose concentrations will be determined by the blood samples taken by ELISA
Changes in blood glucose | day 42
  The glucose concentrations will be determined by the blood samples taken by ELISA
Changes in blood glucose | day 56
  The glucose concentrations will be determined by the blood samples taken by ELISA
Changes in blood glucose | day 70
  The glucose concentrations will be determined by the blood samples taken by ELISA
Changes in blood glucose | day 71
  The glucose concentrations will be determined by the blood samples taken by ELISA
Changes in blood insulin | day 0
  The insulin concentrations will be determined in the blood samples and measured by ELISA
Changes in blood insulin | day 14
  The insulin concentrations will be determined in the blood samples and measured by ELISA
Changes in blood insulin | day 28
  The insulin concentrations will be determined in the blood samples and measured by ELISA
Changes in blood insulin | day 29
  The insulin concentrations will be determined in the blood samples and measured by ELISA
Changes in blood insulin | day 42
  The insulin concentrations will be determined in the blood samples and measured by ELISA
Changes in blood insulin | day 56
  The insulin concentrations will be determined in the blood samples and measured by ELISA
Changes in blood insulin | day 70
  The insulin concentrations will be determined in the blood samples and measured by ELISA
Changes in blood insulin | day 71
  The insulin concentrations will be determined in the blood samples and measured by ELISA
Changes in blood cholesterol | day 0
  The cholesterol concentrations will be determined in the blood samples taken
Changes in blood cholesterol | day 14
  The cholesterol concentrations will be determined in the blood samples taken
Changes in blood cholesterol | day 28
  The cholesterol concentrations will be determined in the blood samples taken
Changes in blood cholesterol | day 29
  The cholesterol concentrations will be determined in the blood samples taken
Changes in blood cholesterol | day 42
  The cholesterol concentrations will be determined in the blood samples taken
Changes in blood cholesterol | day 56
  The cholesterol concentrations will be determined in the blood samples taken
Changes in blood cholesterol | day 70
  The cholesterol concentrations will be determined in the blood samples taken
Changes in blood cholesterol | day 71
  The cholesterol concentrations will be determined in the blood samples taken
Changes in blood triglycerides | day 0
  The triglycerides concentrations will be determined in the blood samples taken
Changes in blood triglycerides | day 14
  The triglycerides concentrations will be determined in the blood samples taken
Changes in blood triglycerides | day 28
  The triglycerides concentrations will be determined in the blood samples taken
Changes in blood triglycerides | day 29
  The triglycerides concentrations will be determined in the blood samples taken
Changes in blood triglycerides | day 42
  The triglycerides concentrations will be determined in the blood samples taken
Changes in blood triglycerides | day 56
  The triglycerides concentrations will be determined in the blood samples taken
Changes in blood triglycerides | day 70
  The triglycerides concentrations will be determined in the blood samples taken
Changes in blood triglycerides | day 71
  The triglycerides concentrations will be determined in the blood samples taken
changes in blood IL-6 | day 0
  The IL-6 concentrations will be determined in the blood samples taken
changes in blood IL-6 | day 14
  The IL-6 concentrations will be determined in the blood samples taken
changes in blood IL-6 | day 28
  The IL-6 concentrations will be determined in the blood samples taken
changes in blood IL-6 | day 29
  The IL-6 concentrations will be determined in the blood samples taken
changes in blood IL-6 | day 42
  The IL-6 concentrations will be determined in the blood samples taken
changes in blood IL-6 | day 56
  The IL-6 concentrations will be determined in the blood samples taken
changes in blood IL-6 | day 70
  The IL-6 concentrations will be determined in the blood samples taken
changes in blood IL-6 | day 71
  The IL-6 concentrations will be determined in the blood samples taken
changes in blood IL-10 | day 0
  The IL-10 concentrations will be determined in the blood samples taken
changes in blood IL-10 | day 14
  The IL-10 concentrations will be determined in the blood samples taken
changes in blood IL-10 | day 28
  The IL-10 concentrations will be determined in the blood samples taken
changes in blood IL-10 | day 29
  The IL-10 concentrations will be determined in the blood samples taken
changes in blood IL-10 | day 42
  The IL-10 concentrations will be determined in the blood samples taken
changes in blood IL-10 | day 56
  The IL-10 concentrations will be determined in the blood samples taken
changes in blood IL-10 | day 70
  The IL-10 concentrations will be determined in the blood samples taken
changes in blood IL-10 | day 71
  The IL-10 concentrations will be determined in the blood samples taken
changes in blood CRP | Day 0
  The CRP concentrations will be determined in the blood samples taken
changes in blood CRP | Day 14
  The CRP concentrations will be determined in the blood samples taken
changes in blood CRP | Day 28
  The CRP concentrations will be determined in the blood samples taken
changes in blood CRP | Day 29
  The CRP concentrations will be determined in the blood samples taken
changes in blood CRP | Day 42
  The CRP concentrations will be determined in the blood samples taken
changes in blood CRP | Day 56
  The CRP concentrations will be determined in the blood samples taken
changes in blood CRP | Day 70
  The CRP concentrations will be determined in the blood samples taken
changes in blood CRP | Day 71
  The CRP concentrations will be determined in the blood samples taken
measure of protein synthesis by isotopic labelling | Day 28
  measurement of protein synthesis using deuterium labelling water
measure of protein synthesis by isotopic labelling | Day 29
  measurement of protein synthesis using deuterium labelling water
measure of protein synthesis by isotopic labelling | Day 70
  measurement of protein synthesis using deuterium labelling water
measure of protein synthesis by isotopic labelling | Day 71
  measurement of protein synthesis using deuterium labelling water
Measure of lipogenesis de novo by isotopic labelling | Day 28
  measurement of lipogenesis using deuterium labelling water
Measure of lipogenesis de novo by isotopic labelling | Day 29
  measurement of lipogenesis using deuterium labelling water
Measure of lipogenesis de novo by isotopic labelling | Day 70
  measurement of lipogenesis using deuterium labelling water
Measure of lipogenesis de novo by isotopic labelling | Day 71
  measurement of lipogenesis using deuterium labelling water
Changes in vascular function | Day 0
  will be determined by measuring minimal and maximal diameter of brachial artery in mm and the percentage of dilatation using the Flow-Mediated Dilatation GE echographer
Changes in vascular function | Day 28
  will be determined by measuring minimal and maximal diameter of brachial artery in mm and the percentage of dilatation using the Flow-Mediated Dilatation GE echographer
Changes in vascular function | Day 42
  will be determined by measuring minimal and maximal diameter of brachial artery in mm and the percentage of dilatation using the Flow-Mediated Dilatation GE echographer
Changes in vascular function | Day 70
  will be determined by measuring minimal and maximal diameter of brachial artery in mm and the percentage of dilatation using the Flow-Mediated Dilatation GE echographer
Changes in microcirculation | Day 0
  will be determined measuring resting state and maximal flow by Flow Laser Doppler Periflux 5000
Changes in microcirculation | Day 28
  will be determined measuring resting state and maximal flow by Flow Laser Doppler Periflux 5000
Changes in microcirculation | Day 42
  will be determined measuring resting state and maximal flow by Flow Laser Doppler Periflux 5000
Changes in microcirculation | Day 70
  will be determined measuring resting state and maximal flow by Flow Laser Doppler Periflux 5000
Changes in mRNA (transcriptomics) derived from Peripheral Blood Monocellular Cells (PBMC) | Day 0
  will be measured by qPCR
Changes in mRNA (transcriptomics) derived from Peripheral Blood Monocellular Cells (PBMC) | Day 14
  will be measured by qPCR
Changes in mRNA (transcriptomics) derived from Peripheral Blood Monocellular Cells (PBMC) | Day 28
  will be measured by qPCR
Changes in mRNA (transcriptomics) derived from Peripheral Blood Monocellular Cells (PBMC) | Day 29
  will be measured by qPCR
Changes in mRNA (transcriptomics) derived from Peripheral Blood Monocellular Cells (PBMC) | Day 42
  will be measured by qPCR
Changes in mRNA (transcriptomics) derived from Peripheral Blood Monocellular Cells (PBMC) | Day 56
  will be measured by qPCR
Changes in mRNA (transcriptomics) derived from Peripheral Blood Monocellular Cells (PBMC) | Day 70
  will be measured by qPCR
Changes in mRNA (transcriptomics) derived from Peripheral Blood Monocellular Cells (PBMC) | Day 71
  will be measured by qPCR
Changes in body composition | Day 0
  will be determined using bioelectric impendence analysis, Quad Scan.
Changes in body composition | Day 28
  will be determined using bioelectric impendence analysis, Quad Scan.
Changes in body composition | Day 42
  will be determined using bioelectric impendence analysis, Quad Scan.
Changes in body composition | Day 70
  will be determined using bioelectric impendence analysis, Quad Scan.
Changes of the microbiota (stool samples) | day 0
  will be determined by the identification of bacterial biodiversity by a genetic sequencing analysis of bacterial DNA
Changes of the microbiota (stool samples) | day 14
  will be determined by the identification of bacterial biodiversity by a genetic sequencing analysis of bacterial DNA
Changes of the microbiota (stool samples) | day 28
  will be determined by the identification of bacterial biodiversity by a genetic sequencing analysis of bacterial DNA
Changes of the microbiota (stool samples) | day 29
  will be determined by the identification of bacterial biodiversity by a genetic sequencing analysis of bacterial DNA
Changes of the microbiota (stool samples) | day 42
  will be determined by the identification of bacterial biodiversity by a genetic sequencing analysis of bacterial DNA
Changes of the microbiota (stool samples) | day 56
  will be determined by the identification of bacterial biodiversity by a genetic sequencing analysis of bacterial DNA
Changes of the microbiota (stool samples) | day 70
  will be determined by the identification of bacterial biodiversity by a genetic sequencing analysis of bacterial DNA
Changes of the microbiota (stool samples) | day 71
  will be determined by the identification of bacterial biodiversity by a genetic sequencing analysis of bacterial DNA
Food statement at inclusion | day 0
  using 3 days food log before day 0

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle Pickering, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Lepine G, Mariotti F, Tremblay-Franco M, Courrent M, Verny MA, David J, Mathe V, Jame P, Anchisi A, Lefranc-Millot C, Perreau C, Guerin-Deremaux L, Chollet C, Castelli F, Chu-Van E, Huneau JF, Remond D, Pickering G, Fouillet H, Polakof S. Increasing plant protein in the diet induces changes in the plasma metabolome that may be beneficial for metabolic health. A randomized crossover study in males. Clin Nutr. 2024 Dec;43(12):146-157. doi: 10.1016/j.clnu.2024.10.009. Epub 2024 Oct 12. PMID 39454458